CLINICAL TRIAL: NCT03149354
Title: Prevalence of Thyroid Function Abnormalities in HIV-infected Patients: State of Play in 2012
Brief Title: Prevalence of Thyroid Function Abnormalities in HIV-infected Patients
Acronym: THYVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2012_843_0013
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Thyroid; HIV Infections
MeSH Terms: conditions — Thyroid Diseases; HIV Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with HIV (Other): Patients with HIV
  Interventions: Other: Assay of TSH, FT3 and FT4 by immuno-radiometric method

INTERVENTIONS:
Other: Assay of TSH, FT3 and FT4 by immuno-radiometric method — Assay of TSH, FT3 and FT4 by immuno-radiometric method Determine the current prevalence of hypothyroidism in HIV-infected patients

SUMMARY:
Review the evolution of thyroid function in HIV-infected patients, with sufficient follow-up.

DETAILED DESCRIPTION:
Since the appearance of high-efficiency anti-retrovirals (HAARTs) in the treatment of Human Immunodeficiency Virus (HIV), several studies have shown an increase in the prevalence of hypothyroidism (frank, rough or low hypothyroidism T4) in cohorts of HIV-infected adults and children. More specifically, rough hypothyroidism (increased TSH and normal thyroid peripheral hormones) have a prevalence of about 3-12% in HIV-treated patients, which is higher than the general population of about 4.3%. The etiology of frustrated hypothyroidism remains debated in the literature; Effects of antiretroviral therapy (ARV) such as Stavudine®, the effect of dyslipidemia, the effect of HIV infection itself, in proportion to severity (expressed as low CD4 cell count) and AIDS stage. Thyroid dysfunction does not appear to be of autoimmune origin, as anti-peroxidase antibodies are rarely present in HIV-infected patients, unlike the general population.

With the increased life expectancy of HIV-infected patients and the indications of different experts to be treated earlier, the duration of exposure to ARVs is also increasing. Therefore, their chronic toxicity deserves particular attention, in particular on thyroid function and / or thyroid hormone metabolism, since iatrogenicity has not been completely ruled out. In addition, clinical evidence suggests that dysthyroids may be corrected or worsened over time in HIV patients (unpublished personal data).

Today, the natural history of frustrated hypothyroidism and its consequences are not reported in patients infected with HIV. However, it is recognized in the elderly, fructified hypothyroidism evolves over time towards frank hypothyroidism; The latter is associated with an increased prevalence of dyslipidemia, atherosclerosis, diastolic hypertension and therefore an increased risk of myocardial infarction.

It therefore seems interesting to review the evolution of thyroid function in HIV-infected patients, with sufficient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Major Patients.
* Infected with HIV, regardless of stage of disease and treatment, diagnosed between January 2001 and December 2012
* Follow-up at the University Hospital of Amiens.

Exclusion Criteria:

* Patients in the THIVY1 study lost to follow-up since 2001, having moved or undergoing therapeutic break-up
* Deceased Patients
* Major protected persons (under guardianship or guardianship)
* Pregnant women
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2012-12-19 (Actual); Primary Completion 2022-12-19 (Estimated); Study Completion 2022-12-19 (Estimated)

PRIMARY OUTCOMES:
Determine the current prevalence of hypothyroidism | 10 years
  Statistical evaluation of the occurrence of hypothyroidism (clinical and frustrated) in HIV-infected patients Presence or absence of hypothyroidism (clinical and frustration) in patients infected with HIV. Hypothyroidism is defined by TSH> 4mUI / ml and / or FT4 <threshold of normal dosage

CONTACTS AND LOCATIONS:
Overall Officials: Rachel DESAILLOUD, PhD, Principal Investigator — CHU AMIENS-PICARDIE
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France